CLINICAL TRIAL: NCT03434067
Title: The Application of Rapid PTH Test Paper in Operation of Hyperparathyroidism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bo Wang,MD (Other)
Responsible Party: Sponsor-Investigator, Bo Wang,MD, Clinical professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: PTH test paper
Record Dates: First submitted 2018-01-27; First posted 2018-02-15 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Hyperthyroidism; Thyroidectomy; PTH; Immunochromatographic
Keywords: hyperthyroidism; thyroidectomy; PTH; immunochromatographic assay
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — In addition to the normal preoperative preparation of blood Biospecimen before admission, the PTH test paper was used to detection the PTH in remanent blood biospecimen .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Primary hyperthyroidism: Patients diagnosed with primary hyperparathyroidism are prepared for parathyroid surgery. PTH test paper is used addtional at the time point according to Miami principle
- Secondary hyperthyroidism: Patients diagnosed with Secondary hyperthyroidism are prepared for parathyroid surgery. PTH test paper is used addtional at the time point according to Miami principle
- Unilateral thyroidectomy: Patients diagnosed with unilateral thyroid benign tumor were prepared for unilateral thyroidectomy. PTH test paper is used addtional at postoperation
- thyroidectomy and bilateral CCD: Patients diagnosed with bilateral thyroid carcinoma were prepared to undergo total thyroidectomy and bilateral central clearing.PTH test paper is used addtional at postoperation

SUMMARY:
The half-life of the parathyroid hormone is about 4min, blood pth test is use in operation to confirm that parathyroid tumor is removed. but the blood pth test is time consuming and unpractical in most of hospital. this study will compare the application of rapid PTH test paper in operation of hyperparathyroidism.PTH test were measured in operation in different way. it will test at the time of preoperation, 15 minutes after surgery, 1 hour after surgery and 24 hours after surgery. thus evaluate the reliability and accuracy of PTH test paper in evaluating the Miami principles with the linear relation of blood PTH and the PTH test paper method.

DETAILED DESCRIPTION:
Primary hyperparathyroidism is a clinically common disease. At present, the gold standard for determining whether the operation is successful is based on the Miami principle. That means The PTH hormone decreased to 30% of the baseline level after 15min after the tumor was removed. However, due to the differences in PTH monitoring conditions in various hospitals, many hospitals cannot perform rapid PTH monitoring in the operation. Therefore many doctors choose rapid freezing pathology to confirm the lesion., This also led to the inability to evaluate PTH in the presence of multiple lesions,and resulting in the need for reoperations.

ELIGIBILITY:
Inclusion Criteria:

* Primary hyperthyroidism.
* Secondary hyperthyroidism
* Unilateral thyroidectomy.
* Total thyroidectomy and bilateral central compartment dissection

Exclusion Criteria:

* age Older than 70 or younger than 18.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We use the characteristics of short half-life of the parathyroid hormone and try to evaluate it by PTH strip semi-quantitative method. PTH, blood calcium and PTH test were measured at pre-operation, 15 minutes after surgery, 1 hour after surgery and 24 hours after surgery. To evaluate the reliability and accuracy of PTH strip in evaluating the Miami principles with the linear relation of blood PTH and the test paper method.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Serum PTH | 0 minutes, 15 minutes, 1 hour and 24 hours post operation
  Routine serum PTH test, using immunoluminescence.
Serum calcium | 0 minutes, 15 minutes, 1 hour and 24 hours post operation
  Routine serum electrolyte detection.
PTH test paper | 0 minutes, 15 minutes, 1 hour and 24 hours post operation
  PTH test paper test for blood

CONTACTS AND LOCATIONS:
Overall Officials: wen-xin zhao, md, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Wen-xin ZHAO, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided